CLINICAL TRIAL: NCT04969380
Title: Safety and Efficacy of Sofacia Treatment to Improve Facial Lines and Wrinkles, to Lift Lax Tissue in the Submental and Neck Zones and to Lift the Eyebrow
Brief Title: SofWave Treatment to Lift Lax Tissue in the Submental and Neck Zones and to Lift the Eyebrow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI IRB HS# 2019-5520
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2021-10

CONDITIONS: Skin Laxity
Keywords: Laxity Brow Lifting Skin Saggy
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- face and/or neck and/or submental zones (Experimental): the full face and/or neck and/or submental zones including 1. -The forehead and temples (left and right including the peri orbital zone) to lift the eyebrows 2. The cheeks (left and right including perioral zone and nasolabial folds) 3. Submental and sides of the neck
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
Eligible patients will receive 2 face and neck treatments (4-6 weeks ± 2 weeks apart) using the SofWave System. Each investigational site would treat the full face and submental zones including 1. The forehead and temples (left and right including the peri orbital zone) to lift the eyebrows 2. The cheeks (left and right including perioral zone and nasolabial folds) 3. Submental and sides of the neck (left and right) to lift lax skin.

All patients will return to the clinic for two follow up visits: 1. 7 days (FU1) post the first treatment (Tx.1). 2. 3 months ± 2 weeks post last treatment (FU2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 35-80.
2. Non-Smoker.
3. Fitzpatrick skin type I-VI.
4. Desire to lift lax skin in the neck and submental and/or to lift the brows.
5. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent
7. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Presence of any active systemic or local infections.
3. Presence of active local skin disease that may alter wound healing.
4. Severe solar elastosis.
5. History of smoking in past 10 years.
6. History of chronic drug or alcohol abuse.
7. Excessive subcutaneous fat on the cheeks.
8. Significant scarring in the area to be treated.
9. Severe or cystic facial acne, acutance uses during past 6 months.
10. Presence of a metal stent or implant in the facial area (dental implants and/or braces are not excluded).
11. Inability to understand the protocol or to give informed consent.
12. History of cosmetic treatments in the facial area to be treated, including facial skin-tightening procedure within the 6 months ; injectable (Botox or fillers) of any type within the 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift, blepharoplasty, or brow lift (including contour threads) within the past 12 months.
13. Taking Isotretinoin or other oral retinoid within the past 6 months; taking anti-platelet or anti-coagulant within the past 2 weeks.
14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Change in lift of lax tissue | 3 and 6 months post last treatment
  As assessed by independent masked evaluators. Quantitative image analysis to objectively measure change in lift of the eyebrow and submental and neck lax tissue would be conducted by comparing baseline images to those taken at each visit post FU1 (Pre Tx.2, FU2)

CONTACTS AND LOCATIONS:
Overall Officials: Ruthie Amir, MD, Study Director — Sofwave
Locations (1):
- University of California, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided